CLINICAL TRIAL: NCT04331327
Title: Clinical and Ultrasonographic Assessment of Effectiveness of Intra-articular Knee Injection Using Platelet Derived Lyophilized Growth Factors in Egyptian Patients With Symptomatic Primary Knee Osteoarthritis
Brief Title: Intra-articular Injection of Allogenic Lyophilized Growth Factors in Primary Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rasmia Elgohary (Other)
Responsible Party: Sponsor-Investigator, Rasmia Elgohary, lecturer of internal medicine, subspecialty rheumatology and clinical immunology, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2016-2017
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Osteo Arthritis Knee
Keywords: osteoarthritis; allogenic platelet rich plasma; lyophilization; growth factors
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic lyophilized growth factors (Active Comparator): Two doses of intra-articular knee injections of lyophilized growth factors were received one dose at the baseline and the other was after 2 months.
  Interventions: Drug: allogenic lyophilized growth factors
- Standard of care (No Intervention): The patients were kept on their traditional medications without any intervention

INTERVENTIONS:
Drug: allogenic lyophilized growth factors — Prior to usage, reconstitution of the product was done using 1-ml saline and 1-ml lignocaine followed by gentle vial rubbing for 3 minutes. Then, the mixture was kept at ambient temperature for 5 minutes to ensure complete protein re-hydration.
  Arms: Allogenic lyophilized growth factors

SUMMARY:
the study was conducted on 31-patients with symptomatic primary knee osteoarthritis. The patients were randomized into intervention and control groups. The control group was kept on their medications without intervention. The intervention group received two doses of allogenic lyophilized growth factors (L-GFs); at baseline and after 2 months.

DETAILED DESCRIPTION:
the study included 31 patients with symptomatic primary knee osteoarthritis (KOA) The study group was randomized into an intervention group and a control one. The control group patients were kept on their traditional medications without any intervention, while intervention group patients were instructed to stop using non-steroidal anti-inflammatory drugs (NSAID) at least 1 week before the assessment and throughout the study. All participants were subjected to baseline clinical, radiographic, and ultrasonography assessment. Follow up assessments was conducted after 6 months.

Patients of the intervention group received two doses of intra-articular knee injections of allogenic lyophilized growth factors (L-GFs); one dose at the baseline and the other was after 2 months.

Lyophilized GFs were prepared at the Cairo Medical Centre Blood Bank from allogenic platelet rich plasma to according a previously published patented method.

Prior to usage, reconstitution of the product was done using 1-ml saline and 1-ml lignocaine followed by gentle vial rubbing for 3 minutes. Then, the mixture was kept at ambient temperature for 5 minutes to ensure complete protein re-hydration.

The injection was done under complete guidance of ultrasonography through lateral supra-patellar short axis in-plane approach under sterile aseptic conditions. After injection, local ice application and oral paracetamol were allowed if the patient felt pain. NSAIDs were completely avoided as they may inhibit the desired post-injection inflammatory process. Patients were encouraged to restrict vigorous knee activities for 48 hours.

ELIGIBILITY:
Inclusion Criteria

* Clinical and radiographic diagnosis of primary knee osteoarthritis
* Patients must be symptomatic

Exclusion Criteria:

* Patients with secondary knee osteoarthritis
* previous intra-articular steroid, or hyaluronic knee injection in last year
* Patients with other disabling lower limb osteoarthropathy or myopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline WOMAC scores at 6 months | At baseline and after 6 months.
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores consist of 24 questions in 3 sections regarding; five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). A sum of the scores for all three sub-scales gives a total WOMAC score. The higher scores mean a worse outcome.
Change from Baseline structural outcomes scores at 6 months | At baseline and after 6 months.
  Knee ultrasonography assessment of effusion, femoral cartilage, anterior horn medial meniscus, synovial hypertrophy

SECONDARY OUTCOMES:
post injection complications of the intervention treatment | at each time following the injection
  The patients of the intervention group were asked if they experienced any adverse events following the injection, with special concern on:
  1. Post-injection pain: Both the duration and intensity were documented. The pain intensity was measured by 0-10 visual analogue scale (VAS).
  2. General symptoms or signs related to infection and allergy such as fever, chills, pruritus, dyspnea, urticaria, or rash.
  3. Erythema, swelling, or abnormal discharge from the site of injection.

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Gado, MD, Principal Investigator — Kasr Alainy School of Medicine, Cairo University
Locations (1):
- rheumatology and clinical immunology unit of internal medicine department of Kasr Al-ainy Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and statistical analysis plan
Supporting Information: Study Protocol, SAP
Time Frame: after publication

REFERENCES:
- [Derived] El-Gohary R, Diab A, El-Gendy H, Fahmy H, Gado KH. Using intra-articular allogenic lyophilized growth factors in primary knee osteoarthritis: a randomized pilot study. Regen Med. 2021 Feb;16(2):113-115. doi: 10.2217/rme-2020-0104. Epub 2021 Mar 23. PMID 33754800
- See also: A patent method describing the preparation of lyophilized growth factors from allogenic platelet rich plasma — https://patentscope.wipo.int/search/en/detail.jsf?docId=WO2018091713